CLINICAL TRIAL: NCT05419947
Title: Randomized Clinical Trial for the Optimization of Indocyanine Green Administration in Near-infrared Fluorescent Cholangiography During Laparoscopic Cholecystectomy.
Brief Title: Clinical Trial for the Optimization of Indocyanine Green Administration in NIRF-C During L.Cholecystectomy.
Acronym: DOTIG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación Instituto de Estudios de Ciencias de la Salud de Castilla y León (Other)
Collaborators: Instituto de Investigación Biomédica de Salamanca (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBS-DOTIG-ECM-2202; 2022-000904-36 (EudraCT Number)
Record Dates: First submitted 2022-05-27; First posted 2022-06-15 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Laparoscopic Cholecystectomy
MeSH Terms: interventions — Solutions; Injections; Indocyanine Green

STUDY DESIGN:
Intervention Model Description: Subjects included in this CT will be treated with VI [Verdye (Diagnostic Green GMBH, Aschheim-Dornach, Germany)]. Single dose and weight-adjusted dose and different administration intervals will be analyzed. Low-intervention clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Fixed dose 3 hours (Experimental): Fixed dose 2.5 mg with IV administration at a time greater than 3 hours before surgery.
  Interventions: Drug: VERDYE powder for solution for injection 25 mg
- Fixed dose 30 min (Experimental): Fixed dose 2.5 mg with IV administration during the immediate preoperative period (15-30 minutes before surgery).
  Interventions: Drug: VERDYE powder for solution for injection 25 mg
- Weight-adjusted dose 3 hour (Experimental): Weight-adjusted dose (0.05 mg/kg of total body weight) with IV administration greater than 3 hours before surgery.
  Interventions: Drug: VERDYE powder for solution for injection 25 mg
- Weight-adjusted dose 30 min (Experimental): Weight-adjusted dose (0.05 mg/kg of total body weight) with IV administration during the immediate preoperative period (15-30 minutes before surgery).
  Interventions: Drug: VERDYE powder for solution for injection 25 mg

INTERVENTIONS:
Drug: VERDYE powder for solution for injection 25 mg — Verdye 25 mg contains sodium VI powder for solution for injection. VI is a water-soluble agent with a spectral absorption peak of 800 nm. It is a drug approved for diagnostic use only and is indicated for the measurement of the excretory function of the liver.
  Other Names: Indocyanine green (ICG)

SUMMARY:
Laparoscopic cholecystectomy is one of the most performed surgical procedures worldwide. One of its most serious complications is injury to the main bile duct, with an incidence of less than 1%. There are different surgical strategies that try to reduce this complication, with indocyanine green fluorescence cholangiography being one of the most recent to appear. This technique is becoming a great tool during laparoscopic cholecystectomy. Despite the great rise of the procedure, today there is a great disparity in the administration protocols of indocyanine green during the procedure.

Goals. The main objective of the study is to analyze whether there are differences between different types of doses and administration intervals of indocyanine green to obtain quality fluorescent cholangiography during laparoscopic cholecystectomy. In addition, the factors that influence the results of the technique will be sought.

DETAILED DESCRIPTION:
Symptomatic cholelithiasis is a pathology of great relevance in the world population, with prevalence rates of up to 20%. The standard treatment for cholelithiasis is laparoscopic cholecystectomy (LC). One of the most serious complications of LC is injury to the main bile duct (LVB). Although this complication has incidences of less than 1% (0.3-0.7% in the different series), the consequences it causes are highly relevant. LVB is related to a significant increase in patient morbidity and mortality, a significant deterioration in quality of life, a very significant increase in healthcare costs and not insignificant medical-legal consequences. Indocyanine green fluorescence cholangiography (CF-VI) is a novel technique that allows precise and real-time anatomical visualization of the extrahepatic biliary anatomy, facilitating surgery and reducing the risk of complications. Currently, there are large differences in LV administration protocols during CF in LC. The precise dose and the ideal moment of administration are key to achieving adequate visualization of the critical vascular and biliary structures and to reduce the fluorescence emitted by the hepatic parenchyma, which could hinder correct anatomical visualization. In relation to the dose, there are many protocols for IV administration, by means of a single dose or a dose adjusted for the patient's body weight. Some authors advocate the administration of IV 24 hours before the procedure, in order to avoid hepatic fluorescence. However, in the context of major outpatient surgery, outpatient surgery or short-stay surgery, we believe that this practice is not currently logistically feasible. Other groups administer the IV with a variable range of time interval. The recent preliminary results of the European Registry of Fluorescent Image Guided Surgery show the great disparity of preoperative LV administration protocols. Therefore, it is necessary to protocolize the administration of the drug based on the results of randomized clinical trials.. The precise dose and the ideal moment of administration are key to achieving adequate visualization of the critical vascular and biliary structures and to reduce the fluorescence emitted by the hepatic parenchyma, which could hinder correct anatomical visualization.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Autonomy, self-sufficiency and independence.
* Scheduled CL indication:
* Symptomatic cholelithiasis: history of biliary colic, acute lithiasic cholecystitis, choledocholithiasis, acute ascending cholangitis of lithiasic origin or acute lithiasic pancreatitis.
* Gallbladder polyps with indication for laparoscopic surgery.
* Vesicular adenomyomatosis with indication for laparoscopic surgery.
* Indication of early LC (<72 hours of admission for acute stone cholecystitis/acute acalculous cholecystitis/complicated biliary colic).
* Deferred urgency LC indication.
* Understanding of information.
* Signature of the informed consent.

Exclusion Criteria:

* Age less than 18 years.
* Disability.
* Pregnancy or lactation.
* Chronic kidney disease (Stage > IIIb).
* Previous adverse reactions or allergies to VI.
* Previous adverse reactions or allergies to VI excipients.
* Adverse reactions or confirmed allergies to iodinated contrast agents.
* Functional thyroid pathology (hyperthyroidism, thyroiditis, toxic multinodular goiter, functioning thyroid adenoma).
* Urgent non-deferrable/emergent gallbladder surgery.
* Initial surgery by laparotomy.
* Previous suspicion of gallbladder carcinoma.
* Inability to understand the information needed to participate in the study.
* Rejection of inclusion within the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime López Sánchez, MD, Principal Investigator — University of Salamanca
Locations (2):
- Spain (2):
  - Hospital Universitario Germans Trias i Pujol., Badalona, Barcelona
  - Complejo Asistencial Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, ICF
Time Frame: From the date of publication of the results.
Access Criteria: Through access to the journal where the results are published.

REFERENCES:
- [Background] Ansaloni L, Pisano M, Coccolini F, Peitzmann AB, Fingerhut A, Catena F, Agresta F, Allegri A, Bailey I, Balogh ZJ, Bendinelli C, Biffl W, Bonavina L, Borzellino G, Brunetti F, Burlew CC, Camapanelli G, Campanile FC, Ceresoli M, Chiara O, Civil I, Coimbra R, De Moya M, Di Saverio S, Fraga GP, Gupta S, Kashuk J, Kelly MD, Koka V, Jeekel H, Latifi R, Leppaniemi A, Maier RV, Marzi I, Moore F, Piazzalunga D, Sakakushev B, Sartelli M, Scalea T, Stahel PF, Taviloglu K, Tugnoli G, Uraneus S, Velmahos GC, Wani I, Weber DG, Viale P, Sugrue M, Ivatury R, Kluger Y, Gurusamy KS, Moore EE. 2016 WSES guidelines on acute calculous cholecystitis. World J Emerg Surg. 2016 Jun 14;11:25. doi: 10.1186/s13017-016-0082-5. eCollection 2016. PMID 27307785
- [Background] Tazuma S, Unno M, Igarashi Y, Inui K, Uchiyama K, Kai M, Tsuyuguchi T, Maguchi H, Mori T, Yamaguchi K, Ryozawa S, Nimura Y, Fujita N, Kubota K, Shoda J, Tabata M, Mine T, Sugano K, Watanabe M, Shimosegawa T. Evidence-based clinical practice guidelines for cholelithiasis 2016. J Gastroenterol. 2017 Mar;52(3):276-300. doi: 10.1007/s00535-016-1289-7. Epub 2016 Dec 10. PMID 27942871
- [Background] Pesce A, Piccolo G, Lecchi F, Fabbri N, Diana M, Feo CV. Fluorescent cholangiography: An up-to-date overview twelve years after the first clinical application. World J Gastroenterol. 2021 Sep 28;27(36):5989-6003. doi: 10.3748/wjg.v27.i36.5989. PMID 34629815
- [Background] Nuzzo G, Giuliante F, Giovannini I, Ardito F, D'Acapito F, Vellone M, Murazio M, Capelli G. Bile duct injury during laparoscopic cholecystectomy: results of an Italian national survey on 56 591 cholecystectomies. Arch Surg. 2005 Oct;140(10):986-92. doi: 10.1001/archsurg.140.10.986. PMID 16230550
- [Background] Strasberg SM, Hertl M, Soper NJ. An analysis of the problem of biliary injury during laparoscopic cholecystectomy. J Am Coll Surg. 1995 Jan;180(1):101-25. No abstract available. PMID 8000648
- [Background] Gupta V, Jain G. Safe laparoscopic cholecystectomy: Adoption of universal culture of safety in cholecystectomy. World J Gastrointest Surg. 2019 Feb 27;11(2):62-84. doi: 10.4240/wjgs.v11.i2.62. PMID 30842813
- [Background] Mascagni P, Vardazaryan A, Alapatt D, Urade T, Emre T, Fiorillo C, Pessaux P, Mutter D, Marescaux J, Costamagna G, Dallemagne B, Padoy N. Artificial Intelligence for Surgical Safety: Automatic Assessment of the Critical View of Safety in Laparoscopic Cholecystectomy Using Deep Learning. Ann Surg. 2022 May 1;275(5):955-961. doi: 10.1097/SLA.0000000000004351. Epub 2020 Nov 16. PMID 33201104
- [Background] Flum DR, Dellinger EP, Cheadle A, Chan L, Koepsell T. Intraoperative cholangiography and risk of common bile duct injury during cholecystectomy. JAMA. 2003 Apr 2;289(13):1639-44. doi: 10.1001/jama.289.13.1639. PMID 12672731
- [Background] Vlek SL, van Dam DA, Rubinstein SM, de Lange-de Klerk ESM, Schoonmade LJ, Tuynman JB, Meijerink WJHJ, Ankersmit M. Biliary tract visualization using near-infrared imaging with indocyanine green during laparoscopic cholecystectomy: results of a systematic review. Surg Endosc. 2017 Jul;31(7):2731-2742. doi: 10.1007/s00464-016-5318-7. Epub 2016 Nov 14. PMID 27844236
- [Background] Ishizawa T, Bandai Y, Ijichi M, Kaneko J, Hasegawa K, Kokudo N. Fluorescent cholangiography illuminating the biliary tree during laparoscopic cholecystectomy. Br J Surg. 2010 Sep;97(9):1369-77. doi: 10.1002/bjs.7125. PMID 20623766
- [Background] Reinhart MB, Huntington CR, Blair LJ, Heniford BT, Augenstein VA. Indocyanine Green: Historical Context, Current Applications, and Future Considerations. Surg Innov. 2016 Apr;23(2):166-75. doi: 10.1177/1553350615604053. Epub 2015 Sep 10. PMID 26359355
- [Background] Lim SH, Tan HTA, Shelat VG. Comparison of indocyanine green dye fluorescent cholangiography with intra-operative cholangiography in laparoscopic cholecystectomy: a meta-analysis. Surg Endosc. 2021 Apr;35(4):1511-1520. doi: 10.1007/s00464-020-08164-5. Epub 2021 Jan 4. PMID 33398590
- [Background] Dip F, LoMenzo E, Sarotto L, Phillips E, Todeschini H, Nahmod M, Alle L, Schneider S, Kaja L, Boni L, Ferraina P, Carus T, Kokudo N, Ishizawa T, Walsh M, Simpfendorfer C, Mayank R, White K, Rosenthal RJ. Randomized Trial of Near-infrared Incisionless Fluorescent Cholangiography. Ann Surg. 2019 Dec;270(6):992-999. doi: 10.1097/SLA.0000000000003178. PMID 30614881
- [Background] van den Bos J, Wieringa FP, Bouvy ND, Stassen LPS. Optimizing the image of fluorescence cholangiography using ICG: a systematic review and ex vivo experiments. Surg Endosc. 2018 Dec;32(12):4820-4832. doi: 10.1007/s00464-018-6233-x. Epub 2018 May 18. PMID 29777357
- [Background] Verbeek FP, Schaafsma BE, Tummers QR, van der Vorst JR, van der Made WJ, Baeten CI, Bonsing BA, Frangioni JV, van de Velde CJ, Vahrmeijer AL, Swijnenburg RJ. Optimization of near-infrared fluorescence cholangiography for open and laparoscopic surgery. Surg Endosc. 2014 Apr;28(4):1076-82. doi: 10.1007/s00464-013-3305-9. PMID 24232054
- [Background] Widjaja SP, Fischer H, Brunner AR, Honigmann P, Metzger J. Acceptance of Ambulatory Laparoscopic Cholecystectomy in Central Switzerland. World J Surg. 2017 Nov;41(11):2731-2734. doi: 10.1007/s00268-017-4098-0. PMID 28660320
- [Background] Agnus V, Pesce A, Boni L, Van Den Bos J, Morales-Conde S, Paganini AM, Quaresima S, Balla A, La Greca G, Plaudis H, Moretto G, Castagnola M, Santi C, Casali L, Tartamella L, Saadi A, Picchetto A, Arezzo A, Marescaux J, Diana M. Fluorescence-based cholangiography: preliminary results from the IHU-IRCAD-EAES EURO-FIGS registry. Surg Endosc. 2020 Sep;34(9):3888-3896. doi: 10.1007/s00464-019-07157-3. Epub 2019 Oct 7. PMID 31591654
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Yokoe M, Hata J, Takada T, Strasberg SM, Asbun HJ, Wakabayashi G, Kozaka K, Endo I, Deziel DJ, Miura F, Okamoto K, Hwang TL, Huang WS, Ker CG, Chen MF, Han HS, Yoon YS, Choi IS, Yoon DS, Noguchi Y, Shikata S, Ukai T, Higuchi R, Gabata T, Mori Y, Iwashita Y, Hibi T, Jagannath P, Jonas E, Liau KH, Dervenis C, Gouma DJ, Cherqui D, Belli G, Garden OJ, Gimenez ME, de Santibanes E, Suzuki K, Umezawa A, Supe AN, Pitt HA, Singh H, Chan ACW, Lau WY, Teoh AYB, Honda G, Sugioka A, Asai K, Gomi H, Itoi T, Kiriyama S, Yoshida M, Mayumi T, Matsumura N, Tokumura H, Kitano S, Hirata K, Inui K, Sumiyama Y, Yamamoto M. Tokyo Guidelines 2018: diagnostic criteria and severity grading of acute cholecystitis (with videos). J Hepatobiliary Pancreat Sci. 2018 Jan;25(1):41-54. doi: 10.1002/jhbp.515. Epub 2018 Jan 9. PMID 29032636
- [Derived] Lopez-Sanchez J, Garrosa-Munoz S, Pardo Aranda F, Gene Skrabec C, Lopez Perez R, Rodriguez-Fortunez P, Sanchez Santos JM, Munoz-Bellvis L; DOTIG Collaborative Group. Dose and administration time of indocyanine green in near-infrared fluorescence cholangiography during laparoscopic cholecystectomy (DOTIG): study protocol for a randomised clinical trial. BMJ Open. 2023 Mar 3;13(3):e067794. doi: 10.1136/bmjopen-2022-067794. PMID 36868593

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The annual rate of LC in the two hospitals in the study is over 300 surgeries per year. In order to recruit 200 in both centres, a review waiting list will be conducted. Patients who meet the inclusion criteria will be given the necessary information and, after signing the informed consent form, will be included in the trial.
Pre-assignment Details: Screening details:
  Patients scheduled for laparoscopic cholecystectomy who meet all inclusion criteria and none of the exclusion criteria
Period: Overall Study
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Started | 49 | 45 | 44 | 62
Completed | 47 | 45 | 44 | 60
Not Completed | 2 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Of the 200 overall number of baseline participants, 196 completed the study; therefore, only the results and data obtained from these 196 subjects were used for the corresponding statistical analyses
Groups:
- Total: Total of all reporting groups
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min | Total
Number analyzed (Participants) | 47 | 45 | 44 | 60 | 196
Age, Customized [Number; unit: participants]
  Between 20 and 91 years | 47 | 45 | 44 | 60 | 200
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Of the 200 overall number of baseline participants, 196 completed the study; therefore, only the results and data obtained from these 196 subjects were used for the corresponding statistical analyses
  Participants
    Female | 33 | 25 | 25 | 38 | 121
    Male | 14 | 20 | 19 | 22 | 75
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Body mass index (BMI) [Mean (Standard Deviation); unit: Kilogram per square meter] | 30.5 (6.3) | 27.1 (4.8) | 28.9 (6.6) | 28.4 (7.1) | 27.9 (8.2)

OUTCOME MEASURES:

1. Primary Outcome: Identification of Biliary Structures Prior to Dissection of the Hepatocystic Triangle.
Description: Identification of biliary structures prior to dissection of the hepatocystic triangle. Participants may be assigned to multiple categories according to the intraoperative identification of distinct anatomical structures observed in each case. The fluorescent green substance, VERDYE, will be injected to the patients in order to visualize the below listed organs once the surgery has begun, but before the disection of the hepatocystic triangle has begun.
  Category 1. Identification of the cystic duct prior to dissection Category 2. Identification of the common bile duct prior to dissection Category 3. Identification of the junction of the cystic duct with the common bile duct prior to dissection Category 4. Identification of the union of the cystic duct with the gallbladder prior to dissection Category 5. Identification of the common hepatic duct prior to dissection Category 6. Identification of biliary anatomical variables prior to dissection
Time Frame: During surgical procedure, before beginning the dissection of the hepatocystic triangle.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  Category 1 | 26 | 20 | 26 | 29
  Category 2 | 32 | 25 | 28 | 36
  Category 3 | 15 | 12 | 18 | 19
  Category 4 | 23 | 19 | 25 | 19
  Category 5 | 16 | 16 | 16 | 25
  Category 6 | 2 | 1 | 1 | 0

2. Primary Outcome: Identification of Biliary Structures After Dissection of the Hepatocystic Triangle.
Description: Identification of biliary structures after dissection of the hepatocystic triangle. Participants may be assigned to multiple categories according to the intraoperative identification of distinct anatomical structures observed in each case. The fluorescent green substance, VERDYE, will be injected to the patients in order to visualize the below listed organs once disection of the hepatocystic triangle has begun.
  Category 1. Identification of the cystic duct prior to dissection Category 2. Identification of the common bile duct prior to dissection Category 3. Identification of the junction of the cystic duct with the common bile duct prior to dissection Category 4. Identification of the union of the cystic duct with the gallbladder prior to dissection Category 5. Identification of the common hepatic duct prior to dissection Category 6. Identification of biliary anatomical variables prior to dissection
Time Frame: During surgical procedure, after dissection of the hepatocystic triangle.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  Category 1 | 40 | 38 | 36 | 45
  Category 2 | 42 | 33 | 35 | 48
  Category 3 | 41 | 35 | 36 | 40
  Category 4 | 41 | 35 | 36 | 40
  Category 5 | 24 | 26 | 25 | 36
  Category 6 | 6 | 5 | 5 | 3

3. Secondary Outcome: Degree of Identification of Biliary Structures Prior to Dissection of the Hepatocystic Triangle.
Description: Degree of identification of biliary structures prior to dissection of the hepatocystic triangle. The fluorescent green substance, VERDYE, will be injected to the patients in order to visualize the below listed organs once the surgery has begun, but before the disection of the hepatocystic triangle has begun.
  The following scale will be used: 1=little, 2=sufficient, 3=quite a bit, 4=good, 5=excellent. It is scale based on the observation of the surgeon, not an international surgical scale. Hence, it does not have a specific name.
Time Frame: During surgical procedure, before beginning the dissection of the hepatocystic triangle.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  1=little | 12 | 20 | 12 | 25
  2=sufficient | 11 | 7 | 4 | 11
  3=quite a bit | 6 | 5 | 9 | 3
  4=good | 11 | 7 | 10 | 13
  5=excellent | 7 | 6 | 9 | 8

4. Secondary Outcome: Degree of Identification of Biliary Structures After Dissection of the Hepatocystic Triangle.
Description: Degree of identification of biliary structures after dissection of the hepatocystic triangle. The fluorescent green substance, VERDYE, will be injected to the patients in order to visualize the below listed organs once the disection of the hepatocystic triangle has begun.
  The following scale will be used: 1=little, 2=sufficient, 3=quite a bit, 4=good, 5=excellent. It is scale based on the observation of the surgeon, not an international surgical scale. Hence, it does not have a specific name.
Time Frame: During surgical procedure, after the disection of the hepatocystic triangle has begun.
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  1=little | 6 | 6 | 5 | 13
  2=sufficient | 6 | 12 | 6 | 10
  3= quite a bit | 8 | 4 | 5 | 5
  4= good | 12 | 6 | 15 | 15
  5= excellent | 15 | 17 | 13 | 17

5. Secondary Outcome: Extent to Which Fluorescence Cholangiography Was Perceived as Useful for Surgery
Description: Extent to which fluorescence cholangiography was perceived as useful for surgery. Participants were assigned toeach category according to the intraoperative identification of distinct anatomical structures observed in each case,once the surgery has begun.
  The following scale will be used: 0=not useful, 1=moderately useful, 2=very useful. It is scale based on the observation of the surgeon, not an international surgical scale. Hence, it does not have a specific name.
Time Frame: During surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  0= not useful | 4 | 9 | 3 | 13
  1= moderately useful | 22 | 24 | 19 | 23
  2= very useful | 21 | 12 | 22 | 24

6. Secondary Outcome: Extent to Which Liver Fundus Fluorescence (Contrast Between Liver and Ducts) Was Perceived as Disturbing.
Description: Extent to which liver fundus fluorescence (contrast between liver and ducts) was perceived as disturbing. Participants were assigned to each category according to the intraoperative identification of distinct anatomical structures observed in each case, once the surgery has begun.
  The following scale will be used: 0=no disturbance, 1=slightly disturbed, 2=disturbed visualization, but cystic-bile duct junction was clearly visible before dissection, 3=disturbed visualization and cystic-bile duct junction was only visible after dissection. dissection and 4= very disturbed: it was impossible to correctly visualize the biliary structures. It is scale based on the observation of the surgeon, not an international surgical scale. Hence, it does not have a specific name.
Time Frame: During surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Fixed Dose 3 Hours | Fixed Dose 30 Min | Weight-adjusted Dose 3 Hour | Weight-adjusted Dose 30 Min
Number analyzed (Participants) | 47 | 45 | 44 | 60
Participants
  Cat 0 | 26 | 12 | 26 | 7
  Cat 1 | 16 | 17 | 13 | 20
  Cat 2 | 4 | 4 | 5 | 15
  Cat 3 | 1 | 9 | 0 | 9
  Cat 4 | 0 | 3 | 0 | 9

ADVERSE EVENTS:
Time Frame: The adverse event collection period in this study extends from the time of surgery until one month postsurgery.
Description: Adverse and serious adverse events were defined per clinical trial guidelines. Events were analyzed collectively, as their occurrence depends on the surgical procedure for each patient's underlying pathology, not on the treatment arm.
Groups:
- Total Number of Patients: All patients who completed the study, regardless of the group to which they were randomized. Adverse events were not analyzed separately by study arm but rather aggregated across all participants. Consequently, in the following sections, all references to adverse events pertain to this combined analysis. This approach was selected because the occurrence of adverse events is primarily related to the surgical intervention required for each patient's underlying pathology, rather than to the treatment arm to which the patient was randomized. Therefore, stratifying adverse events by study arm would not yield specific information regarding the dose or timing of administration of the investigational medicinal product.
Arm/Group | Total Number of Patients
All-Cause Mortality (participants affected / at risk) | 0/196
Serious Adverse Events (participants affected / at risk) | 13/196
Other Adverse Events (participants affected / at risk) | 66/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Number of Patients (N=196)
Adenocarcinoma (Hepatobiliary disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Acute pancreatitis (Gastrointestinal disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Gastrointestinal disorders) | 1 (1)
Cholangitis (Gastrointestinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Intraabdominal fluid collection (Infections and infestations) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Number of Patients (N=196)
Ecchymosis (Vascular disorders) | 2 (2)
Phlebitis (Vascular disorders) | 3 (3)
Haematoma (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Pyrexia (General disorders) | 4 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anxiety disorders (Psychiatric disorders) | 1 (1)
Nervousness (Psychiatric disorders) | 1 (1)
Dehiscense (Injury, poisoning and procedural complications) | 1 (1)
Accident (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 2 (2)
Wound secretion (Injury, poisoning and procedural complications) | 2 (2)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 2 (2)
Headache (Nervous system disorders) | 4 (4)
Disorientation (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (3)
Melaena (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 14 (14)
Acute cholecystitis necrotic (Hepatobiliary disorders) | 1 (1)
Gallbladder rupture (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Omphalitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2)
Sacral pain (Musculoskeletal and connective tissue disorders) | 1 (3)
Abcess (Infections and infestations) | 2 (2)
Abcess intestinal (Infections and infestations) | 2 (2)
Conjunctivitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 3 (3)
Fungal infection (Infections and infestations) | 1 (1)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT05419947/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT05419947/SAP_001.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT05419947/ICF_002.pdf